CLINICAL TRIAL: NCT05635045
Title: A Follow-Up Study to Monitor Therapeutic Response in Transthyretin Cardiac Amyloidosis Using Amyloid Reactive Peptide 124I-evuzamitide (AT01) PET/CT
Brief Title: Evuzamitide in PET/CT to Measure Potential Therapeutic Response in ATTR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Attralus, Inc. (Industry)
Responsible Party: Principal Investigator, Mathew S. Maurer, MD, Arnold and Arlene Goldstein Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAU0561
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Transthyretin Amyloidosis
Keywords: 124I-evuzamitide; Positron Emission Tomography (PET); ATTR-CM
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stabilizer Only (Active Comparator): Subjects treated with tafamidis selected to re-scan to determine the change over time in Evuzamitide uptake
  Interventions: Drug: I 124-Evuzamitide
- Silencer Only (Active Comparator): Subjects treated with vutrisiran selected to re-scan to determine the change over time in Evuzamitide uptake
  Interventions: Drug: I 124-Evuzamitide
- Stabilizer and Silencer (tafamidis + patisiran) (Active Comparator): Subjects treated with tafamidis and patisiran selected to re-scan to determine the change over time in Evuzamitide uptake
  Interventions: Drug: I 124-Evuzamitide
- Stabilizer and Silencer (vutrisiran + diflunisal) (Active Comparator): Subjects treated with vutrisiran and diflunisal selected to re-scan to determine the change over time in Evuzamitide uptake
  Interventions: Drug: I 124-Evuzamitide

INTERVENTIONS:
Drug: I 124-Evuzamitide — Amyloid reactive protein used as imaging agent in whole body SPECT-CT imaging
  Other Names: Attralus AT-01

SUMMARY:
This was a single center, prospective cohort study that is evaluating the ability of 124I-evuzamitide PET scanning to detect potential therapeutic changes in subjects under treatment for ATTR after one year had elapsed since their original 124I-evuzamitide PET scan.

Ten previously scanned subjects re-consented to undergo another 124I-evuzamitide PET scan. Demographic, clinical and phenotypic data were collected to characterize potential changes since their previous scans.

DETAILED DESCRIPTION:
Transthyretin cardiac amyloidosis (ATTR-CA) causes progressive heart disease that is often overlooked. It harms the heart muscle because the unstable, unfurled amyloid proteins fold up into large pieces that get caught in between layers of heart tissue, causing amyloid deposits. The earlier it is detected, the better for the patient.

There is a need to improve the early diagnosis of this disease because echocardiography (sonograms of the heart) and cardiac MRI are not useful enough for this. There is an X-ray of the heart using a compound called PYP that can detect amyloid deposits earlier than ultrasound images or clinical signs, but it's not clear how early it does so. Also, it can't detect amyloid deposits outside the heart, which causes lots of pain and suffering in people with this disease.

In the first phase of this study the radiation compound, evuzamitide, was shown to detect amyloidosis in the heart of selected subjects. So, the investigators used it to detect potential therapeutic changes in 10 subjects undergoing treatment for Transthyretin Amyloidosis.

Changes in the uptake of evuzamitide were compared between subjects treated on stabilizer only, subjects treated on silencer only and subjects treated with two different combinations of stabilizer plus silencer

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
2. Were enrolled in the initial pilot using 124I-Evuzamitide, on ATTR stabilizer and/or silencer therapy. Able to understand and sign the informed consent document after the nature of the study has been fully explained.
3. TTR genotype shown to be either Val122Ile or wild type.

Exclusion Criteria:

Overall Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
2. Were enrolled in the initial pilot using 124I-Evuzamitide, on ATTR stabilizer and/or silencer therapy. Able to understand and sign the informed consent document after the nature of the study has been fully explained.
3. TTR genotype shown to be either Val122Ile or wild type.

The presence of any of the following excludes eligibility for enrollment in this study:

1. Primary amyloidosis (AL) or secondary amyloidosis (AA).
2. Active malignancy or non-amyloid disease with expected survival of less than 1 year.
3. Heart failure, in the opinion of the investigator, primarily caused by something other than amyloidosis.
4. Ventricular assist device.
5. Impairment from stroke, injury or other medical disorder that precludes participation in the study.
6. Disabling dementia or other mental or behavioral disease.
7. Enrollment in a clinical trial not approved for co-enrollment.
8. Continuous intravenous inotropic therapy.
9. Inability or unwillingness to comply with the study requirements.
10. Chronic kidney disease requiring hemodialysis or peritoneal dialysis.
11. Patients taking heparin, or heparin derivatives (e.g. low molecular weight heparins) for anticoagulation.
12. Other reason that would make the subject inappropriate for entry into this study.

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Maurer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smiley DA, Einstein AJ, O'Gorman KJ, Santana D, Teruya S, Chan N, Nalbandian A, Poterucha TJ, Helmke ST, Mintz A, Goldner K, Sekulic M, Mirabal A, Cuomo MO, Guadalupe S, De Los Santos J, Paulino ME, Mateo KA, Rodriguez CM, Jimenez M, Wardhere A, Bampatsias D, Castillo M, Peng B, Maurer MS. Early Detection of Transthyretin Cardiac Amyloidosis Using 124I-Evuzamitide Positron Emission Tomography/Computed Tomography. JACC Cardiovasc Imaging. 2025 Jul;18(7):799-811. doi: 10.1016/j.jcmg.2025.01.018. Epub 2025 May 28. PMID 40439628

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stabilizer Only | Silencer Only | Stabilizer and Silencer (Tafamidis + Patisiran) | Stabilizer and Silencer (Vutrisiran + Diflunisal)
Started | 4 | 1 | 3 | 2
Completed | 4 | 1 | 2 | 2
Not Completed | 0 | 0 | 1 | 0
Not completed — measurements were not usable due material error in imaging agent supplied | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stabilizer Only | Silencer Only | Stabilizer and Silencer (Tafamidis + Patisiran) | Stabilizer and Silencer (Vutrisiran + Diflunisal) | Total
Number analyzed (Participants) | 4 | 1 | 3 | 2 | 10
Age, Continuous [Mean (Full Range); unit: years] | 68.75 [60 to 76] | 65 [65 to 65] | 75 [70 to 80] | 60 [53 to 67] | 67.77 [53 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 4 | 1 | 3 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 1 | 3 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 3 | 0 | 3 | 1 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
TTR Genotype [Count of Participants; unit: Participants]
  Wild-Type | 2 | 0 | 3 | 0 | 5
  V122i | 2 | 0 | 0 | 0 | 2
  Val30Met | 0 | 0 | 0 | 1 | 1
  Thr60Ile | 0 | 1 | 0 | 0 | 1
  Asp38Glu | 0 | 0 | 0 | 1 | 1
PYP Scan result [Count of Participants; unit: Participants] — Grade 0: No myocardial uptake, considered normal. Grade 1: Myocardial uptake is present but less intense than bone (rib) uptake, considered equivocal.
  Grade 2: Myocardial uptake is equal to or greater than bone uptake. Positive for cardiac amyloidosis.
  Grade 3: Myocardial uptake is greater than bone uptake. Strongly positive for cardiac amyloidosis.
  Participants
    PYP Score 0 - no uptake | 0 | 0 | 0 | 0 | 0
    PYP Score 1 - less uptake than bone | 1 | 1 | 0 | 0 | 2
    PYP Score 2 - as much uptake as bone | 0 | 0 | 0 | 1 | 1
    PYP Score 3 - more uptake than bone | 3 | 0 | 2 | 1 | 6
    PYP Score 2 or 3 - indeterminate whether uptake is equal to or greater than bone | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median of Uptake of Evuzamitide as Measured by Volume of Interest in Milliliters
Description: Volumes of interest (VOIs) were manually traced on PET emission images fused with CT images to define the left ventricular (LV) and right ventricular (RV) contours, including cavity blood pool. Blood pool activity concentration was measured in a 10-mm-diameter left atrial spherical VOI. For 124I-evuzamitide, we used a threshold of mean + 2 standard deviations of blood pool activity concentration.
Time Frame: Up to one month after imaging
Population: 1 subject was scanned but their measurements were not usable due material error in imaging agent supplied.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Stabilizer Only | Silencer Only | Stabilizer and Silencer (Tafamidis + Patisiran) | Stabilizer and Silencer (Vutrisiran + Diflunisal)
Number analyzed (Participants) | 4 | 1 | 2 | 2
mL | 78.7 [13.4 to 137.8] | 253.6 [253.6 to 253.6] | 177.2 [-31.2 to 385.5] | 39.6 [1.4 to 77.8]

2. Primary Outcome: Median of Change in Evuzamitide Uptake as Measured by Percentage Change in Injected Dose (%ID)
Description: Median percentage change in injected dose (%ID), calculated as VOI mean activity concentration x VOI volume/injected activity.
Time Frame: Up to one month after imaging
Population: 1 subject was scanned but their measurements were not usable due material error in imaging agent supplied.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Stabilizer Only | Silencer Only | Stabilizer and Silencer (Tafamidis + Patisiran) | Stabilizer and Silencer (Vutrisiran + Diflunisal)
Number analyzed (Participants) | 4 | 1 | 2 | 2
percent change | 0.2 [-0.1 to 0.5] | 0.8 [0.8 to 0.8] | 1.3 [1.2 to 1.5] | 0.3 [0.2 to 0.4]

3. Primary Outcome: Median of Uptake of Evuzamitide as Measured by Cardiac Amyloid Activity (CAA) in Grams
Description: Cardiac amyloid activity (CAA) in grams is measured as VOI mean standardized uptake value times VOI volume. Standardized uptake value was defined as mean or maximal VOI activity concentration/(injected activity/bodyweight), while target-to-background ratio was considered VOI mean activity concentration/blood pool mean activity concentration. VOI volume was manually traced on PET emission images fused with CT images.
Time Frame: Up to one month after imaging
Population: 1 subject was scanned but their measurements were not usable due material error in imaging agent supplied.
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Stabilizer Only | Silencer Only | Stabilizer and Silencer (Tafamidis + Patisiran) | Stabilizer and Silencer (Vutrisiran + Diflunisal)
Number analyzed (Participants) | 4 | 1 | 2 | 2
grams | 180.2 [-75.9 to 437.8] | 852.8 [852.8 to 852.8] | 952.5 [812.5 to 1092.5] | 155.4 [-18.7 to 329.4]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Stabilizer Only | Silencer Only | Stabilizer and Silencer (Tafamidis + Patisiran) | Stabilizer and Silencer (Vutrisiran + Diflunisal)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 1/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stabilizer Only (N=4) | Silencer Only (N=1) | Stabilizer and Silencer (Tafamidis + Patisiran) (N=3) | Stabilizer and Silencer (Vutrisiran + Diflunisal) (N=2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event is listed as known side-effect of agent

LIMITATIONS AND CAVEATS:
Material problems with one dose of agent prevented one subject's measures from being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT05635045/Prot_SAP_000.pdf